CLINICAL TRIAL: NCT00690898
Title: Phase IIIb, Multicentre, Open-label, Single-arm, Study to Assess the Efficacy and Safety of Lanreotide Autogel 120 mg Administered Every 28 Days as Primary Medical Treatment in Acromegalic Patients With Macroadenoma
Brief Title: Lanreotide as Primary Treatment for Acromegalic Patients With Pituitary Gland Macroadenoma
Acronym: PRIMARYS
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Ipsen (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2-79-52030-207; 2007-000155-34 (EudraCT Number); NCT00225134 (obsolete NCT alias)
Record Dates: First submitted 2008-06-03; First posted 2008-06-05 (Estimated); Results first posted 2013-12-23 (Estimated); Last update posted 2022-10-14 (Actual); Status verified 2022-09

CONDITIONS: Acromegaly
MeSH Terms: conditions — Acromegaly

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Lanreotide autogel 120 mg (Experimental)
  Interventions: Drug: Lanreotide autogel 120 mg

INTERVENTIONS:
Drug: Lanreotide autogel 120 mg — 12 months

SUMMARY:
Acromegaly is a chronic disease caused by excessive secretion of growth hormone (GH) and mainly due to benign tumour localized in the pituitary gland.

The disease develops insidiously, causing a gradual progression of symptoms; consequently most patients are diagnosed in their fourth decade of life.

Administration of somatostatin analogues such as lanreotide have been shown to result in normalisation or the decrease of GH and insulin growth factor (IGF-1) levels and improvement of clinical symptoms in acromegalic patients. The purpose of this study is to evaluate whether lanreotide is also effective on tumour volume reduction (tumour shrinkage) and the benefits of this potential tumour shrinkage on disease symptoms and patient's quality of life.

ELIGIBILITY:
Inclusion Criteria:

* The patient has given written informed consent prior to any study related procedures
* The patient is male or female and is aged between 18 and 75 years, inclusive,
* Diagnosis of acromegaly defined by i) GH nadir > 1 ng/mL as assessed by an oral glucose tolerance test for non diabetic patients (central laboratory results) or a mean GH level > 1 ng/mL based on 5 samples taken every 10 to 15 minutes for diabetic patients ( central laboratory results) AND ii) IGF-1 concentrations elevated above the age- and sex-matched normal range for diabetic and non diabetic patients (central laboratory results),
* The patient has a pituitary adenoma with a diameter greater than or equal to 10 mm based on Magnetic Resonance Imaging (MRI) central reading,
* The patient has no visual field defect identified at the visual evaluation, performed by Goldman Visual Fields Analyser and Automated visual field static perimeter, except visual field abnormality at the time of screening and that is in the investigator's Clinical judgement:

  * Not related to the pituitary adenoma
  * Clinically stable condition not presumed to change during the study period
  * Not modifying the ability to evaluate visual field changes related to the macroadenoma

Exclusion Criteria:

* The patient has a history of hypersensitivity to Lanreotide or drugs with a similar chemical structure,
* The patient has received any unlicensed drug within the 30 days prior to the screening visit or is scheduled to receive an unlicensed drug during the course of the study,
* The patient is likely to require treatment during the study with somatostatin analogues other than Lanreotide Autogel 120 mg, dopamine agonist, GH receptor antagonist (pegvisomant), and Cyclosporine or drugs that are not permitted by the study protocol,
* The patient is a female at risk of pregnancy during the study and is not using acceptable contraceptive methods. Females of childbearing potential must provide a negative pregnancy test at start of study and must be using oral, double barrier (condom with spermicidal jelly, foam suppository, or film; diaphragm with spermicide; or male condom and diaphragm with spermicide), injectable contraception or an intra uterine device. Non childbearing potential is defined as post-menopause for at least 1 year, surgical sterilisation or hysterectomy at least three months before the start of the study,
* The patient is pregnant or lactating,
* The patient has a history of, or known current, problems with alcohol abuse,
* The patient has any mental condition rendering the patient unable to understand the nature, scope and possible consequences of the study, and/or evidence of an uncooperative attitude.
* The patient has abnormal baseline findings, any other medical condition(s) or laboratory findings that, in the opinion of the Investigator, might jeopardize the patient's safety or decrease the chance of obtaining satisfactory data needed to achieve the objective(s) of the study,
* The patient has undergone pituitary surgery or pituitary radiotherapy prior to study entry,
* The patient has previously been treated with a somatostatin analogue,
* The patient has received a dopamine agonist or a GH receptor antagonist (pegvisomant) prior to study entry,
* The patient is expected to require pituitary surgery (adenomectomy) or to receive radiotherapy during the study period,
* Patients with suspected associated prolactinoma: prolactin level > 100 ng/mL (central laboratory results),
* Patient is allergic to Gadolinium (MRI contrast agent) or has acute or chronic severe renal insufficiency (glomerular filtration rate <30 mL/min/1.73m2),
* Patient known by Investigator, to have congenital or acquired optic nerve disease or any visual abnormality with risk of worsening during the course of the study (e.g glaucoma), influencing ability to evaluate Visual Field changes related to the macroadenoma.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 108 (Actual)
Dates: Start 2008-05; Primary Completion 2012-02 (Actual); Study Completion 2012-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Ipsen Medical Director, Study Director — Ipsen
Locations (27):
- University Hospital Antwerpen, Edegem, Belgium
- Všeobecná fakultní nemocnice, Karlova Univerzita, Prague, Czechia
- Finland (2):
  - Helsinki University Center Hospital, Helsinki
  - The Turku University Central Hospital, Turku
- France (9):
  - Hopital De Bois Guillaume, Bois-Guillaume
  - CHU Henri Mondor, Créteil
  - CHU Grenoble Albert Michallon, Grenoble
  - CHRU Lille Hopital Claude Huriez, Lille
  - Groupement Hospitalier Est, Lyon
  - Hôpital de la Timone, Marseille
  - Hôpital Bicêtre, Paris
  - Hopital Haut Leveque, Pessac
  - CHU de Reims, Hopital Robert Debré, Reims
- Germany (5):
  - Friedrich-Alexander University, Erlangen
  - Universitatsklinikum Essen, Essen
  - Klinikum der Johann Wolfgang Goethe-Universität, Frankfurt
  - ENDOC Zentrum für Endokrine Tumoren und Praxis für Endokrinologie, Andrologie und medikamentöse Tumortherapie, Hamburg
  - Medizinische Klinik Innenstadt, München
- Italy (3):
  - AOU Policlinico "G. Martino" Messina, Messina
  - Università Federico II di Napoli, Dipartimento di Endocrinologia Molecolare e Clinicae Oncologia, Napoli
  - Università Cattolica del Sacro Cuore, Policlinico A. Gemelli, U.O.C. di Endocrinologia, Roma
- Netherlands (2):
  - ERASMUS MC Rotterdam, Rotterdam
  - UMC Utrecht, Utrecht
- Cerrahpasa Medical Facility, Istanbul, Turkey (Türkiye)
- United Kingdom (3):
  - 27/28 Aberdeen Royal Infirmary, Aberdeen
  - Christie Hospital, Manchester
  - Derriford Hospital, Plymouth

IPD SHARING:
Plan to Share IPD: Yes
Qualified researchers may request access to patient level data and related study documents including the clinical study report, study protocol with any amendments, annotated case report form, statistical analysis plan, and dataset specifications. Patient level data will be anonymized, and study documents will be redacted to protect the privacy of study participants.
  Any requests should be submitted to www.vivli.org for assessment by an independent scientific review board.
Time Frame: Where applicable, data from eligible studies are available 6 months after the studied medicine and indication have been approved in the US and EU or after the primary manuscript describing the results has been accepted for publication, whichever is later.
Access Criteria: Further details on Ipsen's sharing criteria, eligible studies and process for sharing are available here (https://vivli.org/members/ourmembers/).
URL: https://vivli.org/members/ourmembers/

REFERENCES:
- [Result] Caron PJ, Bevan JS, Petersenn S, Flanagan D, Tabarin A, Prevost G, Maisonobe P, Clermont A; PRIMARYS Investigators. Tumor shrinkage with lanreotide Autogel 120 mg as primary therapy in acromegaly: results of a prospective multicenter clinical trial. J Clin Endocrinol Metab. 2014 Apr;99(4):1282-90. doi: 10.1210/jc.2013-3318. Epub 2013 Jan 1. PMID 24423301
- [Derived] Caron PJ, Bevan JS, Petersenn S, Houchard A, Sert C, Webb SM; PRIMARYS Investigators Group. Effects of lanreotide Autogel primary therapy on symptoms and quality-of-life in acromegaly: data from the PRIMARYS study. Pituitary. 2016 Apr;19(2):149-57. doi: 10.1007/s11102-015-0693-y. PMID 26603536

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Newly diagnosed acromegaly patients with pituitary tumour were recruited at 27 investigational sites in 9 countries namely Belgium, Finland, France, Czech Republic, Germany, Italy, the Netherlands, Turkey and the United Kingdom.
Groups:
- Lanreotide Autogel 120 mg: One Lanreotide Autogel subcutaneous (s.c.) injection administered every 28 days for 12 courses as primary medical treatment in newly diagnosed acromegaly patients with pituitary tumour.
Period: SCREENING
Arm/Group | Lanreotide Autogel 120 mg
Started | 108 (Total of patients screened for the study.)
Completed | 90 (Number of patients included in the study.)
Not Completed | 18
Not completed — Screen failure | 18
Period: TREATMENT
Arm/Group | Lanreotide Autogel 120 mg
Started | 90 (Total number of patients treated.)
Completed | 64
Not Completed | 26
Not completed — Adverse Event | 3
Not completed — Lack of Efficacy | 18
Not completed — Withdrawal by Subject | 4
Not completed — Other (not otherwise specified) | 1

BASELINE CHARACTERISTICS:
Arm/Group | Lanreotide Autogel 120 mg
Number analyzed (Participants) | 90
Age, Continuous [Mean (Standard Deviation); unit: years] | 49.5 (12.4)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 47
  Male | 43
Region of Enrollment [Number; unit: participants]
  France | 42
  United Kingdom | 17
  Germany | 10
  Italy | 7
  Netherlands | 4
  Czech Republic | 3
  Finland | 3
  Belgium | 2
  Turkey | 2
Maximum pituitary adenoma diameter (V1) [Mean (Standard Deviation); unit: mm] | 19.0 (7.1)
Acromegaly Symptoms [Mean (Standard Deviation); unit: score on a scale] — Acromegaly symptoms assessed on a scale of 0 to 8 (0- no symptoms to 8-severe/incapacitating).
  score on a scale
    Headache | 2.8 (2.6)
    Excessive perspiration | 4.1 (2.4)
    Fatigue | 4.2 (2.5)
    Soft tissue swelling | 4.1 (2.4)
    Arthralgia | 3.5 (2.6)
Time since acromegaly diagnosis [Mean (Standard Deviation); unit: days] | 121.2 (149.9)
Pituitary gland MRI volume (V1) [Mean (Standard Deviation); unit: mm^3] | 2739.3 (3262.7)
Growth Hormone (GH) level [Mean (Standard Deviation); unit: mcg/L] | 15.0 (18.8)
Insulin-like Growth Factor 1 (IGF-1) level [Mean (Standard Deviation); unit: mcg/L] | 810 (300)
Prolactin level [Mean (Standard Deviation); unit: mcg/L] | 19.0 (20.2)
Global AcroQoL score [Mean (Standard Deviation); unit: score on a scale] — Acromegaly Quality of Life Assessment (AcroQoL) questionnaire response scores range from 0 to 100. Higher scores indicate best possible Quality of Life. AcroQoL not assessed in patients from Turkey and Finland.
  score on a scale | 56.4 (16.1)

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Patients With Relevant Reduction in Pituitary Tumour Volume (as Measured by MRI) From Baseline Volume (Visit 1) to Week 48 (After 12 Injections at Visit 5)
Description: A blinded, centrally assessed evaluation of all MRIs was performed. A 20% reduction from the volume at Visit 1 was considered to be clinically relevant.
Time Frame: Week 1 and Week 48
Population: Analysis based on intent-to-treat (ITT) population comprised of 89 patients.
Measure: Number (95% Confidence Interval); unit: percentage of subjects
Arm/Group | Lanreotide Autogel 120 mg
Number analyzed (Participants) | 89
percentage of subjects
  Greater than or equal to 20% | 62.9 [52.0 to 72.9]
  Less than 20% | 37.1 [27.1 to 48.0]

2. Secondary Outcome: Number of Patients With at Least a 20% Reduction in Tumour Volume From Baseline Volume (Visit 1) to Week 12 (Visit 3) and Week 24 (Visit 4).
Time Frame: Baseline (week 1) to week 12 and week 24
Population: Analysis based on number (n) of subjects in the Intent to Treat population (ITT) with a valid value.
Measure: Number; unit: participants
Arm/Group | Lanreotide Autogel 120 mg
Number analyzed (Participants) | 89
participants
  Greater than or equal to 20% at week 12 (n=85) | 46 [44.7 to 67.3]
  Less than 20% at week 12 (n=85) | 39 [43.0 to 65.0]
  Greater than or equal to 20% at week 24 (n=80) | 45
  Less than 20% at week 24 (n=80) | 35

3. Secondary Outcome: Percent Variation From Baseline to Visit 3, 4 and 5 (Week 12, 24, and 48) of IGF-1 Levels
Time Frame: Week 12, 24, and 48
Population: Analysis based on number (n) of patients with a valid value in the intent-to-treat (ITT) population.
Measure: Mean (95% Confidence Interval); unit: percentage change
Arm/Group | Lanreotide Autogel 120 mg
Number analyzed (Participants) | 89
percentage change
  Week 12 (n=85) | -43.8 [-50.1 to -37.5]
  Week 24 (n=78) | -47.4 [-53.6 to -41.2]
  Week 48 (n=62) | -56.7 [-62.1 to -51.3]

4. Secondary Outcome: Percent Variation From Baseline to Visit 3, 4 and 5 (Week 12, 24, and 48) of Serum GH Levels.
Time Frame: Week 12, 24, and 48
Population: Analysis based on number (n) of subjects in the Intent to Treat population (ITT) with a valid value.
Measure: Mean (95% Confidence Interval); unit: percentage change
Arm/Group | Lanreotide Autogel 120 mg
Number analyzed (Participants) | 85
percentage change
  Week 12 (n=85) | -62.1 [-70.5 to -53.6]
  Week 24 (n=78) | -64.6 [-72.3 to -57.0]
  Week 48 (n=63) | -70.9 [-79.2 to -62.5]

5. Secondary Outcome: Change From Baseline to Visit 3, 4 and 5 (Week 12, 24, and 48) of Prolactin Levels
Time Frame: Week 12, 24 and 48
Population: Analysis based on the number (n) of subjects with baseline level between 20 ng/ml and 100 ng/ml in the ITT population with a valid value.
Measure: Mean (Standard Deviation); unit: mcg/L
Arm/Group | Lanreotide Autogel 120 mg
Number analyzed (Participants) | 21
mcg/L
  Prolactin levels at baseline (n=21) | 48.0 (24.4)
  Change From Baseline to Week 12 (n=20) | -18.0 (19.0) [-26.9 to -9.1]
  Change From Baseline to Week 24 (n=20) | -18.6 (20.3) [-28.1 to -9.1]
  Change From Baseline to Week 48 (n=12) | -17.3 (18.4) [-29.0 to -5.6]

6. Secondary Outcome: Percentage of Patients With Improved, Unchanged or Worsened Clinical Signs of Acromegaly (Arthralgia) From Baseline
Description: The status of clinical signs of acromegaly assessed by an acromegaly symptoms questionnaire (paper form) completed by the patient at each study visit. The scoring for each clinical sign of acromegaly on the questionnaire is from 0 (no symptom) to 8 (severe, incapacitating symptom). The variation (or no variation) in scores indicate whether the clinical sign of acromegaly had improved, worsened or was unchanged.
Time Frame: Week 12, 24 and 48
Population: Analysis based on the number (n) of subjects in the ITT population with a valid value.
Measure: Number; unit: percentage of subjects
Arm/Group | Lanreotide Autogel 120 mg
Number analyzed (Participants) | 89
percentage of subjects
  Baseline to week 12 - Worsened (n=88) | 9.1 [3.1 to 15.1]
  Baseline to week 12 - Unchanged (n=88) | 26.1 [17.0 to 35.3]
  Baseline to week 12 - Improved (n=88) | 64.8 [54.8 to 74.8]
  Baseline to week 24 - Worsened (n=81) | 11.1 [4.3 to 18.0]
  Baseline to week 24 - Unchanged (n=81) | 24.7 [15.3 to 34.1]
  Baseline to week 24 - Improved (n=81) | 64.2 [53.8 to 74.6]
  Baseline to week 48 - Worsened (n=62) | 17.7 [8.2 to 27.3]
  Baseline to week 48 - Unchanged (n=62) | 22.6 [12.2 to 33.0]
  Baseline to week 48 - Improved (n=62) | 59.7 [47.5 to 71.9]

7. Secondary Outcome: Percentage of Patients With Improved, Unchanged or Worsened Clinical Signs of Acromegaly (Excessive Perspiration) From Baseline
Description: as for outcome 6
Time Frame: Week 12, 24 and 48
Population: Analysis based on the number (n) of subjects in the ITT population with a valid value.
Measure: Number; unit: percentage of subjects
Arm/Group | Lanreotide Autogel 120 mg
Number analyzed (Participants) | 88
percentage of subjects
  Baseline to week 12 - Worsened (n=88) | 11.4 [4.7 to 18.0]
  Baseline to week 12 - Unchanged (n=88) | 25.0 [16.0 to 34.0]
  Baseline to week 12 - Improved (n=88) | 63.6 [53.6 to 73.7]
  Baseline to week 24 - Worsened (n=81) | 14.8 [7.1 to 22.6]
  Baseline to week 24 - Unchanged (n=81) | 21.0 [12.1 to 29.9]
  Baseline to week 24 - Improved (n=81) | 64.2 [53.8 to 74.6]
  Baseline to week 48 - Worsened (n=62) | 9.7 [2.3 to 17.0]
  Baseline to week 48 - Unchanged (n=62) | 24.2 [13.5 to 34.9]
  Baseline to week 48 - Improved (n=62) | 66.1 [54.3 to 77.9]

8. Secondary Outcome: Percentage of Patients With Improved, Unchanged or Worsened Clinical Signs of Acromegaly (Fatigue) From Baseline
Description: as for outcome 6
Time Frame: Week 12, 24 and 48
Population: Analysis based on the number (n) of subjects in the ITT population with a valid value.
Measure: Number; unit: percentage of subjects
Arm/Group | Lanreotide Autogel 120 mg
Number analyzed (Participants) | 88
percentage of subjects
  Baseline to week 12 - Worsened (n=88) | 13.6 [6.5 to 20.8]
  Baseline to week 12 - Unchanged (n=88) | 25.0 [16.0 to 34.0]
  Baseline to week 12 - Improved (n=88) | 61.4 [51.2 to 71.5]
  Baseline to week 24 - Worsened (n=81) | 16.0 [8.1 to 24.0]
  Baseline to week 24 - Unchanged (n=81) | 17.3 [9.0 to 25.5]
  Baseline to week 24 - Improved (n=81) | 66.7 [56.4 to 76.9]
  Baseline to week 48 - Worsened (n=62) | 14.5 [5.7 to 23.3]
  Baseline to week 48 - Unchanged (n=62) | 29.0 [17.7 to 40.3]
  Baseline to week 48 - Improved (n=62) | 56.5 [44.1 to 68.8]

9. Secondary Outcome: Percentage of Patients With Improved, Unchanged or Worsened Clinical Signs of Acromegaly (Headache) From Baseline
Description: as for outcome 6
Time Frame: Week 12, 24 and 48
Population: Analysis based on the number (n) of subjects in the ITT population with a valid value.
Measure: Number; unit: percentage of subjects
Arm/Group | Lanreotide Autogel 120 mg
Number analyzed (Participants) | 88
percentage of subjects
  Baseline to week 12 - Worsened (n=88) | 13.6 [6.5 to 20.8]
  Baseline to week 12 - Unchanged (n=88) | 46.6 [36.2 to 57.0]
  Baseline to week 12 - Improved (n=88) | 39.8 [29.5 to 50.0]
  Baseline to week 24 - Worsened (n=81) | 11.1 [4.3 to 18.0]
  Baseline to week 24 - Unchanged (n=81) | 42.0 [31.2 to 52.7]
  Baseline to week 24 - Improved (n=81) | 46.9 [36.0 to 57.8]
  Baseline to week 48 - Worsened (n=62) | 14.5 [5.7 to 23.3]
  Baseline to week 48 - Unchanged (n=62) | 46.8 [34.4 to 59.2]
  Baseline to week 48 - Improved (n=62) | 38.7 [26.6 to 50.8]

10. Secondary Outcome: Percentage of Patients With Improved, Unchanged or Worsened Clinical Signs of Acromegaly (Soft Tissue Swelling) From Baseline
Description: as for outcome 6
Time Frame: Week 12, 24 and 48
Population: Analysis based on the number (n) of subjects in the ITT population with a valid value.
Measure: Number; unit: percentage of subjects
Arm/Group | Lanreotide Autogel 120 mg
Number analyzed (Participants) | 88
percentage of subjects
  Baseline to week 12 - Worsened (n=88) | 10.2 [3.9 to 16.6]
  Baseline to week 12 - Unchanged (n=88) | 26.1 [17.0 to 35.3]
  Baseline to week 12 - Improved (n=88) | 63.6 [53.6 to 73.7]
  Baseline to week 24 - Worsened (n=81) | 11.1 [4.3 to 18.0]
  Baseline to week 24 - Unchanged (n=81) | 22.2 [13.2 to 31.3]
  Baseline to week 24 - Improved (n=81) | 66.7 [56.4 to 76.9]
  Baseline to week 48 - Worsened (n=62) | 14.5 [5.7 to 23.3]
  Baseline to week 48 - Unchanged (n=62) | 19.4 [9.5 to 29.2]
  Baseline to week 48 - Improved (n=62) | 66.1 [54.3 to 77.9]

11. Secondary Outcome: Changes in the Global Acromegaly Quality of Life Assessment (AcroQoL) From Baseline
Description: Acromegaly Quality of Life Assessment (AcroQoL) questionnaire response scores range from 0 to 100. Higher scores indicate best possible Quality of Life.
Time Frame: Week 12, 24 and 48
Population: Analysis based on the number (n) of subjects in the ITT population with a valid value.
Measure: Mean (95% Confidence Interval); unit: units on a scale
Arm/Group | Lanreotide Autogel 120 mg
Number analyzed (Participants) | 84
units on a scale
  Baseline to week 12 (n=82) | 7.8 [5.7 to 9.8]
  Baseline to week 24 (n=75) | 8.0 [5.3 to 10.8]
  Baseline to week 48 (n=59) | 9.5 [6.2 to 12.8]

ADVERSE EVENTS:
Time Frame: Four years
Arm/Group | Lanreotide Autogel 120 mg
Serious Adverse Events (participants affected / at risk) | 13/90
Other Adverse Events (participants affected / at risk) | 72/90
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Lanreotide Autogel 120 mg (N=90)
Anaemia (Blood and lymphatic system disorders) | 1 (1)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Gamma-glutamyltransferase increased (Investigations) | 1 (1)
Hyperparathyroidism (Endocrine disorders) | 1 (1)
Hypophysectomy (Surgical and medical procedures) | 1 (1)
Hypothermia (General disorders) | 1 (1)
Insulin-like growth factor increased (Investigations) | 1 (1)
Intracranial hypotension (Nervous system disorders) | 1 (1)
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 1 (1)
Ovarian cyst (Reproductive system and breast disorders) | 1 (1)
Oxygen saturation decreased (Investigations) | 1 (1)
Pneumoperitoneum (Gastrointestinal disorders) | 1 (1)
Renal colic (Renal and urinary disorders) | 1 (1)
Sleep apnoea syndrome (Respiratory, thoracic and mediastinal disorders) | 1 (2)
Syncope (Nervous system disorders) | 2 (2)
Thyroid cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Thyroid neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Visual acuity reduced (Eye disorders) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Lanreotide Autogel 120 mg (N=90)
Abdominal pain (Gastrointestinal disorders) | 9 (16)
Alopecia (Skin and subcutaneous tissue disorders) | 12 (12)
Cholelithiasis 6 (6.7%) [7] (Hepatobiliary disorders) | 6 (7)
Diarrhoea (Gastrointestinal disorders) | 35 (98)
Fatigue (General disorders) | 5 (5)
Gastrointestinal disorder (Gastrointestinal disorders) | 10 (16)
Nausea (Gastrointestinal disorders) | 6 (14)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No